CLINICAL TRIAL: NCT00992017
Title: A Phase II Study to Assess the Safety and Immunogenicity of an Inactivated Monovalent Influenza A (H1N1) Vaccine in HIV-1 Infected Pregnant Women
Brief Title: Safety of and Immune Response to an H1N1 Influenza Vaccine in HIV Infected Pregnant Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P1086; 10835 (Registry Identifier: DAIDS ES Registry Number); IMPAACT P1086
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Results first posted 2012-03-13 (Estimated); Last update posted 2021-11-05 (Actual); Status verified 2014-12

CONDITIONS: HIV Infections; H1N1 Influenza Virus
Keywords: Vaccine; Pregnant; Perinatal
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- H1N1 vaccine (Experimental): Pregnant women enrolled received two doses of H1N1 vaccine, administered 21 days apart.
  Interventions: Biological: Influenza A (H1N1) monovalent vaccine

INTERVENTIONS:
Biological: Influenza A (H1N1) monovalent vaccine — Two 15-microgram intramuscular vaccine injections given together form one dose; two doses (four total injections) are given 21 days apart

SUMMARY:
Both pregnant women and people infected with HIV are at increased risk of viral infection, including influenza infection. Pregnant women infected with HIV may be at particular risk of infection from the new H1N1 influenza virus. This study tested the safety and immunogenicity of an H1N1 influenza vaccine in pregnant women infected with HIV.

DETAILED DESCRIPTION:
On June 11, 2009, the World Health Organization declared a pandemic of the new H1N1 influenza virus, after the virus had caused significant fevers and respiratory illnesses in Mexico and the United States. Pregnant women are at an increased risk of complications from influenza. HIV infected people tend to have lower than normal antibody responses to seasonal influenza vaccines. Data suggest that larger than average doses of a vaccine counteract a weak antibody response. Preliminary results from ongoing studies of influenza A (H1N1) 2009 monovalent vaccines indicate that the vaccine may increase immune activation. This study tested the safety and antibody response of high doses of the influenza A (H1N1) 2009 monovalent vaccine in pregnant women infected with HIV.

Participation in this study lasted until 6 months after participants had delivered their babies or up to 52 weeks. Participants received two doses of the H1N1 vaccine at study entry and after 21 days. Each dose consisted of two intramuscular injections (four total injections). On the days of the injections, participants had their babies' heart rates checked before and after vaccination. At these visits, and at follow-up visits on Days 21, 31, and 42, participants completed a review of symptoms, physical and neurological exams, and a blood draw. For 10 days after receiving each dose of the vaccine, participants were asked to keep track of their temperatures and symptoms or reactions in a journal. Participants were contacted on Day 2 and Day 10 after the first dose of vaccine was given and on Day 2 after the second dose of vaccine was given. Some participants also received a phone call after 6 months.

At delivery of each participant's baby, blood was drawn from both the mother and umbilical cord (or from the baby if the cord blood could not be obtained). At 3 and 6 months after delivery, participants came in for follow-up visits involving, for both mother and child, a review of symptoms, brief physical exams, and blood draws (at 6 months only some women had a clinic visit, the rest received a phone call).

ELIGIBILITY:
Inclusion Criteria for Step I:

* Confirmed diagnosis of HIV-1 infection
* Pregnant
* Between 14 and 35 weeks of gestation
* Documented platelet count of greater than 50,000 mm3 and an absolute neutrophil count (ANC) of greater than 500 mm3 within 28 days prior to study entry
* Able to understand and comply with planned study procedures
* On antiretroviral therapy (ART) as outlined in the treatment guidelines for pregnant HIV-1 infected women. Women must be currently taking ART or should initiate ART either prior to or concomitantly with the first dose of the vaccine.

Inclusion Criteria for Step II:

* Received the first dose of influenza A (H1N1) 2009 monovalent vaccine
* Has a documented platelet count of greater than 50,000 mm3 and an ANC of greater than 500 mm3 within the 28 days prior to Step II entry

Exclusion Criteria for Step I:

* Has a known allergy to eggs, egg products, neomycin, or polymyxin
* Has a history, in the opinion of the site investigator, of severe reactions following previous immunization with seasonal TIV
* Participation in a novel H1N1 influenza vaccine study in the past 2 years
* Proven history, by reverse transcription polymerase chain reaction (RT-PCR), of novel influenza H1N1 infection or positive influenza diagnostic test since June 2009 (specificity to H1N1 not required) prior to study entry
* Received any other live licensed vaccine within 4 weeks or inactivated licensed vaccine within 2 weeks prior to study entry
* Received a nonlicensed agent (vaccine, drug, biologic, device, blood product, or medication) within 4 weeks prior to vaccination in this study or expects to receive another nonlicensed agent before delivery
* Acute illness and/or an oral temperature greater than or equal to 100.0 degrees F within 24 hours prior to study entry
* Use of anti-cancer chemotherapy or radiation therapy within the preceding 36 months of study enrollment or has immunosuppression as a result of an underlying illness or treatment (other than HIV-1 infection)
* Active neoplastic disease (excluding nonmelanoma skin cancer, human papillomavirus [HPV]-related cervical dysplasia, and cervical intraepithelial neoplasia [CIN] Grades 1, 2, or 3)
* Long-term use of glucocorticoids, including oral or parenteral prednisone or equivalent (at least 2.0 mg/kg per day or at least 20 mg total dose) for more than 2 consecutive weeks (or 2 weeks total) in the past 3 months or high-dose inhaled steroids (more than 800 mcg/day of beclomethasone dipropionate or equivalent) within the past 3 months. Nasal and topical steroids are allowed.
* Received immunoglobulin or other blood products (with exception of Rho D immune globulin) within the 3 months prior to enrollment in this study
* Current diagnosis of uncontrolled major psychiatric disorder
* History of Guillain-Barre syndrome in the subject or subject's family (including parents, siblings, half-siblings, or children)
* Onset of a neurological disorder including (but not limited to) absent ankle and patellar deep tendon reflexes (DTRs) in both legs (all four absent) within the past 6 months
* Disproportionate loss of strength in lower extremity or extremities compared to the upper extremities (not thought to be related to pregnancy) within the past 6 months
* Any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol. Pregnancy complications such as preterm labor, hypertension and pre-eclampsia are not exclusion criteria for this study.

Exclusion Criteria for Step II:

* Received a nonlicensed agent (vaccine, drug, biologic, device, blood product, or medication), other than from participation in this study, since the study vaccine dose #1 or expects to receive another nonlicensed agent before delivery
* Use of anti-cancer chemotherapy or radiation therapy since study vaccine dose #1, new diagnosis of an active malignancy, or is immunosuppressed as a result of an underlying illness (other than HIV-1 infection) or treatment
* Use of glucocorticoids, including oral or parenteral prednisone or equivalent (at least 2.0 mg/kg per day or at least 20 mg total dose) or high-dose inhaled steroids (more than 800 mcg/day of beclomethasone dipropionate or equivalent) for more than 2 consecutive weeks (or 2 weeks total) since study vaccine dose #1. Nasal and topical steroids are allowed.
* Received immunoglobulin or other blood products (with exception of Rho D immune globulin) since study vaccine dose #1
* A new diagnosis of uncontrolled major psychiatric disorder since study vaccine dose #1
* New occurrence or new awareness of Guillain-Barre syndrome in the subject or subject's family (including parents, siblings, half-siblings, or children) since study vaccine dose #1
* A new onset of a neurological disorder including (but not limited to) absent ankle and patellar DTRs in both legs (all four absent) since study vaccine dose #1
* Disproportionate loss of strength in lower extremity or extremities compared to the upper extremities (not thought to be related to pregnancy) since study vaccine dose #1
* Any Grade 3 toxicity or AE experienced by a participant unless the investigator has received protocol team approval
* Any Grade 4 toxicity or AE (other than injection site reaction or fever) that is definitely, probably, or possibly related to the study vaccine dose #1
* Any Grade 4 injection site reactions or fever experienced by a subject, unless the investigator has received protocol team approval
* Any Grade 4 AEs that are definitely not or probably not related to study vaccine, unless the investigator has received protocol team approval
* Any new clinical findings since the study vaccine dose #1, that, in the investigator's opinion, would compromise the safety of the participant
* Participant refuses further vaccination. The subject will still be asked to complete safety visits and be followed in the study.
* Participant withdraws consent. Participants may withdraw their consent for study participation at any time and for any reason, without penalty.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2009-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Nachman, MD, Study Chair — State University of New York at Stony Brook
Locations (31):
- United States (29):
  - Usc La Nichd Crs, Alhambra, California
  - University of California, UC San Diego CRS, La Jolla, California
  - Miller Children's Hosp. Long Beach CA NICHD CRS, Long Beach, California
  - UCLA-Los Angeles/Brazil AIDS Consortium (LABAC) CRS, Los Angeles, California
  - Univ. of California San Francisco NICHD CRS, San Francisco, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Washington Hosp. Ctr. NICHD CRS, Washington D.C., District of Columbia
  - South Florida CDTC Ft Lauderdale NICHD CRS, Fort Lauderdale, Florida
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Pediatric Perinatal HIV Clinical Trials Unit CRS, Miami, Florida
  - USF - Tampa NICHD CRS, Tampa, Florida
  - Rush Univ. Cook County Hosp. Chicago NICHD CRS, Chicago, Illinois
  - Ann & Robert H. Lurie Children's Hospital of Chicago (LCH) CRS, Chicago, Illinois
  - Tulane Univ. New Orleans NICHD CRS, New Orleans, Louisiana
  - Johns Hopkins Univ. Baltimore NICHD CRS, Baltimore, Maryland
  - Children's Hosp. of Boston NICHD CRS, Boston, Massachusetts
  - Boston Medical Center Ped. HIV Program NICHD CRS, Boston, Massachusetts
  - WNE Maternal Pediatric Adolescent AIDS CRS, Worcester, Massachusetts
  - Rutgers - New Jersey Medical School CRS, Newark, New Jersey
  - Metropolitan Hosp. NICHD CRS, New York, New York
  - Columbia IMPAACT CRS, New York, New York
  - SUNY Stony Brook NICHD CRS, Stony Brook, New York
  - Bronx-Lebanon CRS, The Bronx, New York
  - Jacobi Med. Ctr. Bronx NICHD CRS, The Bronx, New York
  - DUMC Ped. CRS, Durham, North Carolina
  - The Children's Hosp. of Philadelphia IMPAACT CRS, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital CRS, Memphis, Tennessee
  - Texas Children's Hospital CRS, Houston, Texas
  - Seattle Children's Research Institute CRS, Seattle, Washington
- Puerto Rico (2):
  - University of Puerto Rico Pediatric HIV/AIDS Research Program CRS, San Juan
  - San Juan City Hosp. PR NICHD CRS, San Juan

REFERENCES:
- [Background] Novel Swine-Origin Influenza A (H1N1) Virus Investigation Team; Dawood FS, Jain S, Finelli L, Shaw MW, Lindstrom S, Garten RJ, Gubareva LV, Xu X, Bridges CB, Uyeki TM. Emergence of a novel swine-origin influenza A (H1N1) virus in humans. N Engl J Med. 2009 Jun 18;360(25):2605-15. doi: 10.1056/NEJMoa0903810. Epub 2009 May 7. PMID 19423869
- [Background] Jamieson DJ, Honein MA, Rasmussen SA, Williams JL, Swerdlow DL, Biggerstaff MS, Lindstrom S, Louie JK, Christ CM, Bohm SR, Fonseca VP, Ritger KA, Kuhles DJ, Eggers P, Bruce H, Davidson HA, Lutterloh E, Harris ML, Burke C, Cocoros N, Finelli L, MacFarlane KF, Shu B, Olsen SJ; Novel Influenza A (H1N1) Pregnancy Working Group. H1N1 2009 influenza virus infection during pregnancy in the USA. Lancet. 2009 Aug 8;374(9688):451-8. doi: 10.1016/S0140-6736(09)61304-0. Epub 2009 Jul 28. PMID 19643469
- [Result] S. Nachman, A. Weinberg, P. Muresan, M. Abzug, R. Ebiasah, E. Petzold, B. Heckman, H. Watts, J. Miller and M. Levin Safety of an Inactivated Influenza A (H1N1) 2009 Monovalent Vaccine (H1N1 vaccine) in HIV-1 Infected Pregnant Women, P1086. Presented at the Retroviruses Conference, Feb 2010
- [Result] Weinberg A, Muresan P, Fenton T, Handelsman E, Watts H, Miller J, Heckman B, Bloom A, Ebiasah R, Petzold E, Levy W, Abzug M, Levin M and Nachman S for IMPAACT P1086 Team: Safety and Immunogenicity of Two Doses of Monovalent Pandemic H1N1 (pH1N1) Influenza Vaccine in HIV-Infected Pregnant Women. Presented at the IDSA conference, October 2010.
- [Derived] Abzug MJ, Nachman SA, Muresan P, Handelsman E, Watts DH, Fenton T, Heckman B, Petzold E, Weinberg A, Levin MJ; International Maternal Pediatric Adolescent AIDS Clinical Trials Group P1086 Protocol Team. Safety and immunogenicity of 2009 pH1N1 vaccination in HIV-infected pregnant women. Clin Infect Dis. 2013 May;56(10):1488-97. doi: 10.1093/cid/cit057. Epub 2013 Feb 1. PMID 23378284
- See also: Click here for information on the IMPAACT group and for the package insert on the H1N1 vaccine. — http://www.impaactgroup.org
- See also: Click here for the table used for grading toxicities: DAIDS Grading Severity of AEs, V1.0, Dec04 — http://rsc.tech-res.com/safetyandpharmacovigilance/gradingtables.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pregnant women were enrolled from 31 sites between October 8, 2009 and November 13, 2009.
Pre-assignment Details: Two study participants were enrolled but left the clinic before receiving any vaccination and they were taken off study.
Groups:
- H1N1 Vaccine: Pregnant women received two doses of H1N1 vaccine administered 21 days apart. Each dose consisted of two 15-microgram intramuscular injections.
Period: Overall Study
Arm/Group | H1N1 Vaccine
Started | 128 (Two additional women were enrolled but left the clinic before vaccine was administered.)
Received Both Study Vaccinations | 124
Received Only One Study Vaccination | 4 (Reasons: delivered and LFU; moved; no transportation; ineligible - blood transfusion at delivery)
Completed | 118
Not Completed | 10
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 2
Not completed — Unable to get to clinic | 5
Not completed — Not adhere to study requirements | 1

BASELINE CHARACTERISTICS:
Arm/Group | H1N1 Vaccine
Number analyzed (Participants) | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 112
  Puerto Rico | 16
CD4 Cells Count [Mean (Standard Deviation); unit: cells / mm^3] — This measures the number of CD4 cells.
  cells / mm^3 | 504 (264)
Percentage of CD4 Cells [Mean (Standard Deviation); unit: percentage of CD4 cells] — This measures the percentage of CD4 cells.
  percentage of CD4 cells | 30 (11)
Gestational Age [Mean (Standard Deviation); unit: Weeks] — This shows the approximate gestational age at study entry.
  Weeks | 25 (6)

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Who Had at Least One Adverse Event (AE)
Description: Shows the number of participants who had at least one adverse event (AE) in each category. These include: abnormal laboratory values, signs and symptoms, or diagnoses; solicited local AEs; and solicited systemic AEs. Adverse Events were graded using the DAIDS Grading Severity of AEs (see Link under More Information), as follows: grade 1=mild, 2=moderate, 3=severe, 4=life threatening/disabling, 5=death.
Time Frame: Measured up to 6 months after delivery
Population: All 128 pregnant women who received at least one vaccination are included in this analysis.
Measure: Number; unit: Participants
Groups:
- H1N1 Vaccine: Pregnant women enrolled in the study.
Arm/Group | H1N1 Vaccine
Number analyzed (Participants) | 128
Participants
  Overall (New AEs after start of treatment) | 118
  Grade 4 AEs (New, after start of treatment) | 11
  Grade 3 AEs (New, after start of treatment) | 8
  Grade >=2 local and systemic AEs to injection | 0

2. Primary Outcome: The Number of Participants Who Had at Least One AE Attributed to the Study Vaccine
Description: Shows the number of participants who experienced any events that were thought to be at least possibly related to study treatment. Adverse Events were graded using the DAIDS Grading Severity of AEs (see Link under More Information), as follows: grade 1=mild, 2=moderate, 3=severe, 4=life threatening/disabling, 5=death.
Time Frame: Measured up to 6 months after delivery
Population: All 128 pregnant women who received at least one vaccination are included.
Measure: Number; unit: Participants
Groups:
- Vaccinated Study Participants: Pregnant women who received at least one H1N1 vaccination.
Arm/Group | Vaccinated Study Participants
Number analyzed (Participants) | 128
Participants | 0

3. Primary Outcome: Withholding of Second Vaccine Dose Due to Adverse Reactions Attributed to First Dose
Time Frame: Measured at Day 21
Population: All 128 pregnant women who received at least one vaccination are included.
Measure: Number; unit: Participants
Arm/Group | Vaccinated Study Participants
Number analyzed (Participants) | 128
Participants | 0

4. Primary Outcome: Percent of Pregnant Women With a Hemagglutination Inhibition (HAI) Titer of >= 40
Description: Antibodies to Influenza A (H1N1) 2009 were measured using an HAI assay. The potential titer read-outs from the assay used were <10 (considered undetectable), 10, 20, 40, 60, 80, 160, 320, 640, and >=1280. Seroprotection was defined as having a titer of >=40 following vaccination.
Time Frame: Measured at 21 days after first dose and at 10 days after second dose of study vaccine
Population: The analysis population consists of the eligible pregnant women with nonmissing HAI titers, who had not delivered prior to the evaluation, and had received all doses of vaccine up to that timepoint. The N for the analyses of HAI titers after the first and second vaccinations were 118 and 108, respectively.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Groups:
- H1N1 Vaccine: The pregnant women who received the H1N1 vaccinations.
Arm/Group | H1N1 Vaccine
Number analyzed (Participants) | 118
Percent of participants
  Percent with titers >= 40 post dose 1 (N=118) | 73.7 [64.8 to 81.4]
  Percent with titers >= 40 post dose 2 (N=108) | 80.6 [71.8 to 87.5]

5. Secondary Outcome: Percent of Pregnant Women With an HAI Titer of >= 40 at Delivery, 3 Months and 6 Months After Delivery
Description: as for outcome 4
Time Frame: Measured at delivery of the baby, and at 3 months and 6 months after delivery
Population: The population consists of eligible pregnant women with nonmissing HAI titers, who had not delivered before the evaluation post second dose, and received two doses of vaccine. The N for the analyses of HAI titers at delivery, and at 3 and 6 months after were 102, 92 and 58, respectively. Only some women had a clinic visit at 6 months post delivery.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Groups:
- H1N1 Vaccine: Pregnant women who received H1N1 vaccinations.
Arm/Group | H1N1 Vaccine
Number analyzed (Participants) | 102
Percent of participants
  % with titers >= 1:40 at delivery (N=102) | 65.7 [55.6 to 74.8]
  % with titers >= 1:40 at 3 mo post delivery (N=92) | 55.4 [44.7 to 65.8]
  % with titers >= 1:40 at 6 mo post delivery (N=58) | 60.3 [46.6 to 73.0]

6. Secondary Outcome: Percent of Infants With an HAI Titer of >= 40
Description: as for outcome 4
Time Frame: Measured at birth (via cord blood) and at 3 months and 6 months of age
Population: The population consists of infants born to eligible women with nonmissing HAI titers, who had not delivered before the evaluation post second dose, and received two doses of vaccine. The N for analyses at birth, 3 and 6 months were 96, 87 and 52, respectively. Cord blood was used when available. Only some infants had a clinic visit at 6 months.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Groups:
- Infants: Infants born to pregnant women who received H1N1 vaccines.
Arm/Group | Infants
Number analyzed (Participants) | 96
Percent of participants
  % infants with titers >= 1:40 at birth (N=96) | 64.6 [54.2 to 74.1]
  % infants with titers >= 1:40 at 3 months (N=87) | 23.0 [14.6 to 33.2]
  % infants with titers >= 1:40 at 6 months (N=52) | 11.5 [4.4 to 23.4]

7. Secondary Outcome: Maternal Geometric Mean Titers (GMT) of Antibodies HAI
Description: Presents the value of the geometric mean titer at each time point. Antibodies to Influenza A (H1N1) 2009 were measured using an HAI assay. The potential titer read-outs from the assay used were <10 (considered undetectable), 10, 20, 40, 60, 80, 160, 320, 640, and >=1280.
Time Frame: Measured after the first and second doses of the vaccine, at delivery, and at 3 and 6 months after delivery
Population: The population consists of eligible women with nonmissing HAI titers, who had not delivered before the evaluation post first or second dose, and received all vaccines up to that point, respectively. The N for analyses after the first and second vaccinations, at delivery, 3 and 6 months after were 104, 94, 102, 92 and 58, respectively.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Groups:
- H1N1 Vaccine: Pregnant women who received the H1N1 vaccines.
Arm/Group | H1N1 Vaccine
Number analyzed (Participants) | 104
titers
  Post first vaccination (N=104) | 83 [63 to 110]
  Post second vaccination (N=94) | 81 [62 to 106]
  At delivery (N=102) | 50 [39 to 65]
  At 3 months post delivery (N=92) | 36 [28 to 46]
  At 6 months post delivery (N=58) | 38 [29 to 50]

8. Secondary Outcome: Infant GMT of Antibodies HAI
Description: as for outcome 7
Time Frame: Measured at birth and at 3 and 6 months of age
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: units on the HAI titer scale
Arm/Group | Infants
Number analyzed (Participants) | 96
units on the HAI titer scale
  At birth (N=96 infants) | 56 [43 to 72]
  At 3 months (N=87 infants) | 13 [11 to 16]
  At 6 months (N=52 infants) | 14 [11 to 17]

9. Secondary Outcome: Maternal Cell-mediated Immunity (CMI) Responses, as Measured by B-cell and T-cell Enzyme-linked Immunosorbent Spot (ELISPOT) Assay Values
Description: The median and interquartile range (IQR) of B-Cell ELISPOT-measured IgG antibody-secreting cells (ASC)/10^6 PBMC and the median and interquartile range (IQR) of T-Cell ELISPOT-measured pH1N1 IFNgamma spot-forming cells (SFC)/10^6 PBMC.
Time Frame: Measured at entry, at 21 days after first dose of vaccine, at 10 days after second dose
Population: The pregnant women who had not delivered prior to the evaluation, had received all doses of vaccine up to that timepoint and had sufficient samples for testing.
Measure: Median (Inter-Quartile Range); unit: ASC or SFC/10^6 PBMC
Arm/Group | H1N1 Vaccine
Number analyzed (Participants) | 45
ASC or SFC/10^6 PBMC
  IgG ASC/10^6 PBMC, Week 0 (N=36) | 6 [2 to 28]
  IgG ASC/10^6 PBMC, Post Dose 1 (N=36) | 15 [4 to 46]
  IgG ASC/10^6 PBMC, Post Dose 2 (N=39) | 14 [6 to 70]
  pH1N1 IFNgamma SFC/10^6 PBMC, Week 0 (N=45) | 166 [38 to 324]
  pH1N1 IFNgamma SFC/10^6 PBMC, Post Dose 1 (N=44) | 117 [40 to 506]
  pH1N1 IFNgamma SFC/10^6 PBMC, Post Dose 2 (N=43) | 76 [32 to 336]

10. Secondary Outcome: Response to Seasonal Trivalent Influenza Vaccine (TIV)
Description: Presents the value of the median titer as well as the interquartile range at study entry. Antibodies to seasonal Influenza vaccine were measured using an HAI assay. The potential titer read-outs from the assay used were <10 (considered undetectable), 10, 20, 40, 60, 80, 160, 320, 640, and >=1280.
Time Frame: Measured at entry
Population: Pregnant women who received the first H1N1 immunization.
Measure: Median (Inter-Quartile Range); unit: titer
Arm/Group | H1N1 Vaccine
Number analyzed (Participants) | 128
titer | 20 [10 to 40]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the date of enrollment in the study until 6 months after delivery.
Description: Include Adverse Events (AEs) of All Grades, Including Abnormal Laboratory Values, Signs and Symptoms, or Diagnoses; Solicited Local AEs and Systemic AEs. Adverse Events were graded using the DAIDS Grading Severity of AEs (see Link under More Information), as follows: grade 1=mild, 2=moderate, 3=severe, 4=life threatening/disabling, 5=death.
Arm/Group | H1N1 Vaccine
Serious Adverse Events (participants affected / at risk) | 21/128
Other Adverse Events (participants affected / at risk) | 118/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | H1N1 Vaccine (N=128)
Vomiting (Gastrointestinal disorders) | 1
Influenza like illness (General disorders) | 1
Pneumonia (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
VIIth nerve paralysis (Nervous system disorders) | 1
Complication of pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 1
Placenta accreta (Pregnancy, puerperium and perinatal conditions) | 1
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 5
Premature labour (Pregnancy, puerperium and perinatal conditions) | 3
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 1
Conversion disorder (Psychiatric disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | H1N1 Vaccine (N=128)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 9
Abdominal pain (Gastrointestinal disorders) | 12
Diarrhoea (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 24
Vomiting (Gastrointestinal disorders) | 15
Fatigue (General disorders) | 9
Pyrexia (General disorders) | 8
Bacterial disease carrier (Infections and infestations) | 7
Vaginitis bacterial (Infections and infestations) | 8
Vulvovaginal candidiasis (Infections and infestations) | 16
Alanine aminotransferase increased (Investigations) | 10
Aspartate aminotransferase increased (Investigations) | 8
Blood albumin abnormal (Investigations) | 30
Blood alkaline phosphatase increased (Investigations) | 7
Blood bicarbonate abnormal (Investigations) | 14
Blood glucose decreased (Investigations) | 16
Blood sodium decreased (Investigations) | 25
Haemoglobin decreased (Investigations) | 21
Back pain (Musculoskeletal and connective tissue disorders) | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11
Dizziness (Nervous system disorders) | 9
Headache (Nervous system disorders) | 31
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 7
Vaginal discharge (Reproductive system and breast disorders) | 19
Vaginal haemorrhage (Reproductive system and breast disorders) | 9
Vulvovaginal pruritus (Reproductive system and breast disorders) | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 22
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 18
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11
Rash (Skin and subcutaneous tissue disorders) | 7
Hypertension (Vascular disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No